CLINICAL TRIAL: NCT03696056
Title: Improving Cognition in Breast Cancer Survivors Using Meditation: A Pilot Study
Brief Title: Improving Brain Function After Breast Cancer Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Ashley M. Henneghan, Assistant Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018-05-0155
Record Dates: First submitted 2018-09-29; First posted 2018-10-04 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Breast Cancer Survivors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kirtan Kriya meditation (Experimental): Participants will mediate for 12 minutes a day for 8 consecutive weeks.
  Interventions: Behavioral: Kirtan Kriya meditation
- Relaxing instrumental music (Active Comparator): Participants will relax listening to music for 12 minutes a day for 8 consecutive weeks.
  Interventions: Behavioral: Music listening program

INTERVENTIONS:
Behavioral: Kirtan Kriya meditation — The program incorporates song with visualization and mudras, and is a multi-faceted, multisensory exercise that appears to engage several areas of the brain implicated in cognitive decline, yet is simple to learn and practice. The meditation includes a repeated Kirtan or song, a mudra or physical/motor component, and a visualization component. The meditation sound file will contain a user friendly introduction to the Kirtan Kriya meditation technique along with detailed instructions and meditation tracks. Three tracks will contain 12 minute guided meditations with the same female voice, and 2 with nature sounds, 2 without any additional sounds. Another 2 tracks will provide only the timing cues (1 with nature sounds, 1 without) so that the participant can conduct the meditation session without guidance if they chose.
  Arms: Kirtan Kriya meditation
Behavioral: Music listening program — The participants will receive audio files and an instruction sheet to facilitate their practice.
  The audio tracks are 12 minutes in length and contain relaxing instrumental music from Mozart, Bach, Beethoven, Debussy, and Pachebel. Participants are instructed to sit comfortably with their eyes closed and listen to a track of their choice for 12 min daily, for 8 weeks and to record each session on their practice log.
  Arms: Relaxing instrumental music

SUMMARY:
This study will explore the feasibility and potential effects of a simple, home-based daily meditation intervention on breast cancer survivors' cognitive and psychological functioning as well as inflammatory regulation.

DETAILED DESCRIPTION:
This study will compare two home based 8-week interventions (Kirtan Kriya meditation vs.

relaxing instrumental music listening) in 40 breast cancer survivors ages 21-75 who completed chemotherapy 3 months to 5 years prior.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a history of non-inflammatory breast cancer (stages I-IV):
* Received chemotherapy as part of their treatment
* Completed chemotherapy treatment 3 months to 10 years prior to study enrollment
* Individuals who have report cognitive deficits

Exclusion Criteria:

* Breast cancer survivors with a history of metastases to the brain
* A physician diagnosis of: dementia, a learning disability, unmanaged major depression, psychosis, schizophrenia, bipolar, traumatic brain injury, cancer of the central nervous system, diabetes, arthritis
* Taking oral steroids within 30 days of enrolling
* A regular meditation practice (greater than 1 time per week)
* Currently taking immune modifying medications

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Verbal learning and memory performance-Hopkins Verbal Learning Test Immediate and Delayed Recall | Baseline, Time 2 (8 weeks after baseline), and Time 3 (16 weeks after baseline).
  The change of the Hopkins Verbal Learning Test-Revised scores for immediate and delayed recall from baseline to Time 3 (16 weeks after baseline) will be assessed. This test measures immediate and delayed verbal memory. Measured as words recalled and adjusted for age and education. Higher words recalled suggests greater verbal learning and memory performance.
Verbal Fluency Performance-Controlled Oral Word Association Test | Baseline, Time 2 (8 weeks after baseline), and Time 3 (16 weeks after baseline).
  The change of the Controlled Oral Word Association Test, a measure of verbal fluency, scores from baseline to Time 3 (16 weeks after baseline) will be assessed. Measured as number of words produced and adjusted for age and education. Higher words produced suggests greater verbal fluency performance.
Executive Functioning Performance- Trail Making Test Parts A & B | Baseline, Time 2 (8 weeks after baseline), and Time 3 (16 weeks after baseline).
  The change in Trails A & B scores, a measure of processing speed and executive attention, from baseline to Time 3 (16 weeks after baseline) will be assessed. Where time until completion is measured and adjusted for age and education. Faster time until completion suggests higher executive function.

SECONDARY OUTCOMES:
Granulocyte-macrophage colony-stimulating factor concentration | Baseline, and Time 2 (8 weeks after baseline).
  The change of concentration in picograms per millilitre from will be assessed baseline to Time 2 (8 weeks after baseline).
Interferon gamma concentration | Baseline, and Time 2 (8 weeks after baseline).
  The change of concentration in picograms per millilitre from baseline to Time 2 (8 weeks after baseline) will be assessed.
Interleukin-1 β concentration | Baseline, and Time 2 (8 weeks after baseline).
  The change of concentration in picograms per millilitre from baseline to Time 2 (8 weeks after baseline) will be assessed.
Interleukin-2 concentration | Baseline, and Time 2 (8 weeks after baseline).
  The change of concentration in picograms per millilitre from baseline to Time 2 (8 weeks after baseline) will be assessed.
Interleukin-4 concentration | Baseline, and Time 2 (8 weeks after baseline).
  The change of concentration in picograms per millilitre from baseline to Time 2 (8 weeks after baseline) will be assessed.
Interleukin-5 concentration | Baseline, and Time 2 (8 weeks after baseline).
  The change of concentration in picograms per millilitre from baseline to Time 2 (8 weeks after baseline) will be assessed.
Interleukin-6 concentration | Baseline, and Time 2 (8 weeks after baseline).
  The change of concentration in picograms per millilitre from baseline to Time 2 (8 weeks after baseline) will be assessed.
Interleukin-7 concentration | Baseline, and Time 2 (8 weeks after baseline).
  The change of concentration in picograms per millilitre from baseline to Time 2 (8 weeks after baseline) will be assessed.
Interleukin-8 concentration | Baseline, and Time 2 (8 weeks after baseline).
  The change of concentration in picograms per millilitre from baseline to Time 2 (8 weeks after baseline) will be assessed.
Interleukin-10 concentration | Baseline, and Time 2 (8 weeks after baseline).
  The change of concentration in picograms per millilitre from baseline to Time 2 (8 weeks after baseline) will be assessed.
Interleukin-12 concentration | Baseline, and Time 2 (8 weeks after baseline).
  The change of concentration in picograms per millilitre from baseline to Time 2 (8 weeks after baseline) will be assessed.
Interleukin-13 concentration | Baseline, and Time 2 (8 weeks after baseline).
  The change of concentration in picograms per millilitre from baseline to Time 2 (8 weeks after baseline) will be assessed.
Tumor necrosis factor alpha concentration | Baseline, and Time 2 (8 weeks after baseline).
  The change of concentration in picograms per millilitre from baseline to Time 2 (8 weeks after baseline) will be assessed.
Self-reported cognitive function | Baseline, Time 2 (8 weeks after baseline), and Time 3 (16 weeks after baseline).
  The change of Functional Assessment of Cancer Therapy-Cognitive for perceived cognitive function and impact on quality of life from baseline to Time 3 (16 weeks after baseline) will be assessed. Lower scores indicate worse functioning. This scale demonstrated adequate reliability in our previous study (Cronbach's α 0.98).
Anxiety Symptoms | Baseline, Time 2 (8 weeks after baseline), and Time 3 (16 weeks after baseline).
  The changes of anxiety symptoms will be assessed with the Patient-Reported Outcomes Measurement Information System scale from baseline to Time 3 (16 weeks after baseline).
  The Patient-Reported Outcomes Measurement Information System (PROMIS) scale will be used to measure anxiety Short Form 8a. Higher scores indicate greater anxiety. This scale demonstrated adequate reliability in our previous study (Cronbach's α's 0.96).
Feelings of depression | Baseline, Time 2 (8 weeks after baseline), and Time 3 (16 weeks after baseline).
  The changes of feelings of depression will be assessed with the Patient-Reported Outcomes Measurement Information System scale from baseline to Time 3 (16 weeks after baseline).
  The Patient-Reported Outcomes Measurement Information System (PROMIS) scale will be used to measure depressive symptoms using the Short Form 8a. This 10-item scale measures the degree that life circumstances are appraised as having been stressful in the previous 4 weeks. Higher scores indicate greater feeling of depression. This scale demonstrated adequate reliability in our previous study (Cronbach's α's 0.96).
Perceived Fatigue | Baseline, Time 2 (8 weeks after baseline), and Time 3 (16 weeks after baseline).
  The changes of fatigue symptoms will be assessed with the Patient-Reported Outcomes Measurement Information System scale from baseline to Time 3 (16 weeks after baseline). The PROMIS Fatigue- Short Form 8a will be used to evaluate fatigue. Higher scores indicate greater fatigue. This measure demonstrated adequate reliability in our previous study (Cronbach's α 0.93).
Perceived stress | Baseline, Time 2 (8 weeks after baseline), and Time 3 (16 weeks after baseline).
  The changes in perceived stress will be assessed with the Perceived Stress Scale from baseline to Time 3 (16 weeks after baseline). Measures the perception of stress with a 10 item scale. Higher scores indicate greater perceived stress.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Only group averaged data will be presented and published.

REFERENCES:
- [Derived] Henneghan AM, Becker H, Harrison ML, Inselmann K, Fico B, Schafer H, King E, Patt D, Kesler S. A randomized control trial of meditation compared to music listening to improve cognitive function for breast cancer survivors: Feasibility and acceptability. Complement Ther Clin Pract. 2020 Nov;41:101228. doi: 10.1016/j.ctcp.2020.101228. Epub 2020 Sep 11. PMID 32949954